CLINICAL TRIAL: NCT07225634
Title: An Open Label, Pharmacokinetic and Safety Study of Combogesic® IV in Pediatric Patients With Acute Pain
Brief Title: A Study of Combogesic® IV (Intravenous) in Pediatric Patients With Acute Pain
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AFT Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFT-MXIV-08p
Record Dates: First submitted 2025-10-30; First posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Ibuprofen; Solutions

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combogesic® IV (Experimental): Combogesic® IV (acetaminophen 10 mg/ml + ibuprofen 3 mg/ml in 100 ml solution for infusion), will be administered by injection into a dedicated indwelling venous cannula, infused over 15 minutes every 6 hours
  Interventions: Drug: Combogesic® IV (fixed-dose combination containing acetaminophen 10 mg/ml + ibuprofen 3 mg/ml in 100 ml solution for infusion)

INTERVENTIONS:
Drug: Combogesic® IV (fixed-dose combination containing acetaminophen 10 mg/ml + ibuprofen 3 mg/ml in 100 ml solution for infusion) — Acetaminophen 1000 mg and Ibuprofen 300 mg per 100 mL solution for intravenous infusion administered as a 15-minute infusion, every 6 hours, as necessary.

SUMMARY:
Combogesic® IV is an intravenous medicine (given by vein) containing a combination of two pain relief (analgesic) medicines called ibuprofen and acetaminophen. The goal of this clinical trial is to study the way that the body processes and clears the intravenous infusion of Combogesic® IV and that it is safe to be used in children and adolescents between the ages of 2 and <17 years.

What will the study involve for participants?

* Combogesic® IV will be administered every 6 hours as necessary with a maximum of 4 doses within a 24-hour period as an intravenous infusion for about 15 minutes.
* Participants will receive Combogesic® IV for a minimum of 12 hours (2 doses) up to a maximum of 5 days (20 doses). Dosing will be dependent on body weight.
* If pain is not sufficiently controlled by Combogesic® IV, opioids may be used as supplementary pain relief at the discretion of the study doctor.
* Have their blood samples collected before dosing and at specific times after dosing. The amount of study drug in the blood will be measured, and safety assessments (including blood and urine samples) will be done.
* Rate the study drug at the end of the treatment.

It is expected that Combogesic® IV will be well tolerated in children and adolescents and that the pharmacokinetics findings will be similar as compared with adults.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female aged between 2 and <17 years.
2. Have a clinical indication of acute pain* requiring hospitalization and multiple doses of parenterally administered nonopioid analgesic medication for at least 0.5 - 5 days.
3. Is either able to provide written informed consent or consent is provided from parents/legal guardians and assent provided from participants (where appropriate).
4. Is willing and able to remain at the study site for at least 12 hours and to attend a follow-up visit at 7 ± 2 days after the last dose of study drug.
5. Have negative HIV and hepatitis B & C test results.

   * Acute pain indications may include but are not limited to post-operative pain associated with musculoskeletal or soft tissue surgery, fractures or injury, or medical procedures.

Exclusion Criteria:

1. Has a known history of allergic reaction or clinically significant intolerance to acetaminophen, aspirin, opioids, or any nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen); history of NSAID-induced bronchospasm (subjects with the triad of asthma, nasal polyps, and chronic rhinitis are at greater risk for bronchospasm and should be considered carefully); or hypersensitivity, allergy, or significant reaction to sulfa (including sulfonamide) medicines, ingredients of the study drug, or any other drugs used in the study including anesthetics and antibiotics that may be required.
2. Has experienced any surgical complications or other issues that, in the opinion of the Investigator, could compromise the safety of the subject if he or she participates in the study or could confound the results of the study.
3. Has any clinically significant unstable cardiac, respiratory, neurological, immunological, hematological, or renal disease or any other condition that, in the opinion of the Investigator, could compromise the subject's welfare, ability to communicate with the study staff, or otherwise contraindicate study participation.
4. Has a history or current diagnosis of a significant psychiatric disorder that, in the opinion of the Investigator, would affect the subject's ability to comply with the study requirements.
5. Has a history of a clinically significant (Investigator opinion) gastrointestinal (GI) event within 6 months before screening or has any history of peptic or gastric ulcers or GI bleeding.
6. Has a surgical or medical condition of the GI or renal system that might significantly alter the absorption, distribution, or excretion of any drug substance.
7. Is considered by the Investigator, for any reason to be an unsuitable candidate to receive the study drug.
8. Is receiving systemic chemotherapy, has an active malignancy of any type, or has been diagnosed with cancer within 5 years before Screening (excluding treated squamous or basal cell carcinoma of the skin).
9. Is currently receiving anticoagulants (e.g. heparin or warfarin).
10. Has received a course of systemic corticosteroids (either oral or parenteral) within 3 months before screening (inhaled nasal steroids and regional/limited area application of topical corticosteroids (Investigator discretion) are allowed).
11. Has a history of chronic use (defined as daily use for > 2 weeks) of NSAIDs, opiates, or glucocorticoids (except inhaled nasal steroids and regional/limited topical corticosteroids), for any condition within 6 months before study drug administration. Aspirin at a daily dose of ≤ 325 mg is allowed for cardiovascular prophylaxis if the subject has been on a stable dose regimen for ≥ 30 days before screening and has not experienced any relevant medical problem.
12. Has a significant renal or hepatic disease, as indicated by clinical laboratory assessment (results ≥ 3 times the upper limit of normal [ULN] for any liver function test, including aspartate aminotransferase [AST], alanine aminotransferase [ALT], or creatinine ≥ 1.5 times the ULN).
13. Has any clinically significant laboratory finding at screening that, in the opinion of the Investigator, contraindicates study participation.
14. Participated in another clinical study within 30 days before Screening.
15. Pregnant or lactating females
16. Sexually active females of childbearing potential not using adequate contraception** and sexually active males not using adequate contraception* **Methods of contraception that are deemed adequate have failure rates of < 1%, including: established use of oral contraceptives in conjunction with a barrier method of contraception; injected or implanted hormonal methods of contraception; placement of intrauterine device (IUD) or intrauterine system (IUS); sexual abstinence; hysterectomy; post-menopausal; sterilized; vasectomy. Suitable contraception should be used for the entire study period, from screening to follow-up. Women of childbearing age include all women that have begun puberty and had their first menstrual period until they reach menopause.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The incidence of treatment-emergent adverse events (TEAEs) associated with exposure to Combogesic® IV in pediatric patients | From start of exposure to Combogesic® IV up to 7 days after last dose
  TEAEs occurring at any timepoint during the treatment period will be coded to MedDRA System Organ Class Code and Preferred Term and tabulated as frequencies and percentages.

SECONDARY OUTCOMES:
The time course of treatment-emergent adverse events | From start of exposure to Combogesic® IV up to 7 days after last dose
The incidence of treatment-related adverse events | From start of exposure to Combogesic® IV up to 7 days after last dose
The incidence of treatment-emergent adverse events of interest (cardiovascular, gastrointestinal, renal, hepatic, administration site conditions and bleeding-related events) | From start of exposure to Combogesic® IV up to 7 days after last dose
Changes in heart rate | From baseline up to 7 days after last dose of Combogesic® IV
Changes in biochemistry values (Aspartate transaminase) | From baseline up to 7 days after last dose
  The number of cases with normal baseline laboratory tests changed to abnormal at the end of the treatment period, and abnormal baseline laboratory tests worsened at the end of the treatment period, with the severity of changes summarized as proportional effects will be evaluated.
Patient's global evaluation of the study drug | From Day 1 until completion of treatment period up to 5 days.
  Each patient will rate the study medication using a questionnaire of:
  How do you rate the study medication?
  1. = Poor;
  2. = Fair;
  3. = Good;
  4. = Very Good;
  5. = Excellent
  The patient's global evaluation of the study drug will be summarized by the number and percentage of subjects within each category.
Define the pharmacokinetic parameters of Combogesic® IV (Cmax - Maximum measured plasma concentration) | Pre-dose of Combogesic® IV to 6 hours post infusion
  This will be estimated for paracetamol and ibuprofen from the plasma concentration against time data, using a non-compartmental model
Consumption of supplemental opioid medication in each 24-hour period as Morphine Milligram Equivalent (MME). | From start of exposure to Combogesic® IV until up to 5 days
Define the pharmacokinetic parameters of Combogesic® IV (Tmax - Time of maximum measured plasma concentration) | Pre-dose of Combogesic® IV to 6 hours post infusion
  This will be estimated for paracetamol and ibuprofen from the plasma concentration against time data, using a non-compartmental model
Define the pharmacokinetic parameters of Combogesic® IV ( t½ - Time required for the plasma drug concentration to decrease by one half) | Pre-dose of Combogesic® IV to 6 hours post infusion
  This will be estimated for paracetamol and ibuprofen from the plasma concentration against time data, using a non-compartmental model
Define the pharmacokinetic parameters of Combogesic® IV (AUC(0-t) - The area under the plasma concentration versus time curve from time zero to the last measurable concentration) | Pre-dose of Combogesic® IV to 6 hours post infusion
  This will be estimated for paracetamol and ibuprofen from the plasma concentration against time data, using a non-compartmental model
Define the pharmacokinetic parameters of Combogesic® IV (Extrapolated AUC(0-∞)- The area under the plasma concentration versus time curve, from zero to infinity) | Pre-dose of Combogesic® IV to 6 hours post infusion
  This will be estimated for paracetamol and ibuprofen from the plasma concentration against time data, using a non-compartmental model
Changes in blood pressure | From baseline up to 7 days after last dose of Combogesic® IV
Changes in body temperature | From baseline up to 7 days after last dose of Combogesic® IV
Changes in respiratory rate | From baseline up to 7 days after last dose of Combogesic® IV
Changes in hematology values (Hemaglobin) | From baseline up to 7 days after last dose
  The number of cases with normal baseline laboratory tests changed to abnormal at the end of the treatment period, and abnormal baseline laboratory tests worsened at the end of the treatment period, with the severity of changes summarized as proportional effects will be evaluated.
Changes in hematology values (Hematocrit) | From baseline up to 7 days after last dose
  The number of cases with normal baseline laboratory tests changed to abnormal at the end of the treatment period, and abnormal baseline laboratory tests worsened at the end of the treatment period, with the severity of changes summarized as proportional effects will be evaluated.
Changes in hematology values (Platelet count) | From baseline up to 7 days after last dose
  The number of cases with normal baseline laboratory tests changed to abnormal at the end of the treatment period, and abnormal baseline laboratory tests worsened at the end of the treatment period, with the severity of changes summarized as proportional effects will be evaluated.
Changes in hematology values (Red Blood Cell (RBC) count) | From baseline up to 7 days after last dose
  The number of cases with normal baseline laboratory tests changed to abnormal at the end of the treatment period, and abnormal baseline laboratory tests worsened at the end of the treatment period, with the severity of changes summarized as proportional effects will be evaluated.
Changes in hematology values (White Blood Cell (WBC) count) | From baseline up to 7 days after last dose
  The number of cases with normal baseline laboratory tests changed to abnormal at the end of the treatment period, and abnormal baseline laboratory tests worsened at the end of the treatment
Changes in hematology values (Differential Leukocyte Count (DLC)) | From baseline up to 7 days after last dose
  The number of cases with normal baseline laboratory tests changed to abnormal at the end of the treatment period, and abnormal baseline laboratory tests worsened at the end of the treatment period, with the severity of changes summarized as proportional effects will be evaluated.
Changes in biochemistry values (Sodium) | From baseline up to 7 days after last dose
  The number of cases with normal baseline laboratory tests changed to abnormal at the end of the treatment period, and abnormal baseline laboratory tests worsened at the end of the treatment period, with the severity of changes summarized as proportional effects will be evaluated.
Changes in biochemistry values (Potassium) | From baseline up to 7 days after last dose
  The number of cases with normal baseline laboratory tests changed to abnormal at the end of the treatment period, and abnormal baseline laboratory tests worsened at the end of the treatment period, with the severity of changes summarized as proportional effects will be evaluated.
Changes in biochemistry values (Urea) | From baseline up to 7 days after last dose
  The number of cases with normal baseline laboratory tests changed to abnormal at the end of the treatment period, and abnormal baseline laboratory tests worsened at the end of the treatment period, with the severity of changes summarized as proportional effects will be evaluated.
Changes in biochemistry values (Creatinine) | From baseline up to 7 days after last dose
  The number of cases with normal baseline laboratory tests changed to abnormal at the end of the treatment period, and abnormal baseline laboratory tests worsened at the end of the treatment period, with the severity of changes summarized as proportional effects will be evaluated.
Changes in biochemistry values (Phosphate) | From baseline up to 7 days after last dose
  The number of cases with normal baseline laboratory tests changed to abnormal at the end of the treatment period, and abnormal baseline laboratory tests worsened at the end of the treatment period, with the severity of changes summarized as proportional effects will be evaluated.
Changes in biochemistry values (Glucose) | From baseline up to 7 days after last dose
  The number of cases with normal baseline laboratory tests changed to abnormal at the end of the treatment period, and abnormal baseline laboratory tests worsened at the end of the treatment period, with the severity of changes summarized as proportional effects will be evaluated.
Changes in biochemistry values (Albumin) | From baseline up to 7 days after last dose
  The number of cases with normal baseline laboratory tests changed to abnormal at the end of the treatment period, and abnormal baseline laboratory tests worsened at the end of the treatment period, with the severity of changes summarized as proportional effects will be evaluated.
Changes in biochemistry values (Total protein) | From baseline up to 7 days after last dose
  The number of cases with normal baseline laboratory tests changed to abnormal at the end of the treatment period, and abnormal baseline laboratory tests worsened at the end of the treatment period, with the severity of changes summarized as proportional effects will be evaluated.
Changes in biochemistry values (Alkaline phosphates) | From baseline up to 7 days after last dose
  The number of cases with normal baseline laboratory tests changed to abnormal at the end of the treatment period, and abnormal baseline laboratory tests worsened at the end of the treatment period, with the severity of changes summarized as proportional effects will be evaluated.
Changes in biochemistry values (Gamma-glutamyl transferase) | From baseline up to 7 days after last dose
  The number of cases with normal baseline laboratory tests changed to abnormal at the end of the treatment period, and abnormal baseline laboratory tests worsened at the end of the treatment period, with the severity of changes summarized as proportional effects will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours Children's Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No